CLINICAL TRIAL: NCT00810862
Title: A 3-Week, Single-Blind, Placebo-Controlled, Within-Patient, Randomized Study of Pimecrolimus Treatment for Atopic Dermatitis of African American Children
Brief Title: Study of Pimecrolimus Treatment for Atopic Dermatitis of African American Children
Status: Terminated | Phase: Phase 4 | Type: Interventional
Why Stopped: Lack of subject enrollment over the past two years.
Sponsor: Children's Hospital of Michigan (Other)
Collaborators: Novartis Pharmaceuticals (Industry)
Responsible Party: Paul J Munzenberger Pharm D Associate Professor, Children's Hospital of Michigan
Allocation: Randomized | Model: Single Group | Masking: Single | Purpose: Treatment
Other Study IDs: pimecrolimus1
Record Dates: First submitted 2008-12-17; First posted 2008-12-18 (Estimated); Last update posted 2008-12-18 (Estimated); Status verified 2008-12

CONDITIONS: Atopic Dermatitis
Keywords: African American children
MeSH Terms: conditions — Dermatitis, Atopic | interventions — pimecrolimus

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Pimecrolimus (Experimental): Pimecrolimus 1% cream
  Interventions: Drug: pimecrolimus active cream
- 2 (Placebo Comparator): Placebo cream over affected study area
  Interventions: Other: placebo base cream

INTERVENTIONS:
Drug: pimecrolimus active cream — Pimecrolimus 1% cream apply to affected study area twice daily for 21 days
  Other Names: Elidel 1% cream Novartis Pharmaceuticals
  Arms: Pimecrolimus
Other: placebo base cream — apply to affected study area twice daily for 21 days
  Other Names: Elidel base cream without active agent; by Novartis Pharmaceuticals
  Arms: 2

SUMMARY:
Primecrolimus cream 1% is effective in the treatment of atopic dermatitis in African American children.

ELIGIBILITY:
Inclusion Criteria:

* African American children aged 2 to 17 years
* mild to moderate atopic dermatitis

Exclusion Criteria:

* m-EASI less than 3 at baseline
* allergy to Elidel or components
* use of oral steroids, immunosuppressive agents,cytostatics of phototherapy within 4 weeks prior to study.
* previous continuous or non-continuous use of pimecrolimus or tacrolimus for greater than 11 months within 2 weeks of enrollment.
* active skin infections.
* immunocompromised patients.
* previous history of skin cancer or lymphoma
* any hypopigmentation in study areas
* pregnant or breastfeeding
* participation in another investigational trial

Ages: 2 Years to 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 18 (Actual)
Dates: Start 2006-11; Primary Completion 2008-06 (Actual); Study Completion 2008-06 (Actual)

PRIMARY OUTCOMES:
Mean change in modified Modified EASI score a dermatologic evaluation of response to topical therapy for atopic dermatitis | at baseline, one week and three weeks following treatment initiation

SECONDARY OUTCOMES:
modified IGA score | at baseline, one week and three weeks following initiation of therapy
hypopigmentation scale score | baseline, one and three weeks following initiation of treatment